CLINICAL TRIAL: NCT04287686
Title: A Randomized, Open Label, Controlled Clinical Study to Evaluate the Recombinant Human Angiotensin-converting Enzyme 2 (rhACE2) in Adult Patients With COVID-19
Brief Title: Recombinant Human Angiotensin-converting Enzyme 2 (rhACE2) as a Treatment for Patients With COVID-19
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Without CDE Approval
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Yimin LI, Director Physician, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIRH-APN01
Record Dates: First submitted 2020-02-21; First posted 2020-02-27 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; Renin-angiotensin-system (RAS)
MeSH Terms: conditions — COVID-19 | interventions — alunacedase alfa

STUDY DESIGN:
Intervention Model Description: 2-arm pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rhACE2 group (Experimental): 0.4 mg/kg IV BID for 7 days (unblinded) + standard of care
  Interventions: Drug: Recombinant human angiotensin-converting enzyme 2 (rhACE2)
- Control group (No Intervention): Standard of care; no placebo

INTERVENTIONS:
Drug: Recombinant human angiotensin-converting enzyme 2 (rhACE2) — In this study, the experimental group will receive 0.4 mg/kg rhACE2 IV BID for 7 days.
  Arms: rhACE2 group

SUMMARY:
This is an open label, randomized, controlled, pilot clinical study in patients with COVID-19, to obtain preliminary biologic, physiologic, and clinical data in patients with COVID-19 treated with rhACE2 or control patients, to help determine whether a subsequent Phase 2B trial is warranted.

DETAILED DESCRIPTION:
This is a small pilot study investigating whether there is any efficacy signal that warrants a larger Phase 2B trial, or any harm that suggests that such a trial should not be done. It is not expected to produce statistically significant results in the major endpoints. The investigators will examine all of the biologic, physiological, and clinical data to determine whether a Phase 2B trial is warranted.

Primary efficacy analysis will be carried only on patients receiving at least 4 doses of active drug. Safety analysis will be carried out on all patients receiving at least one dose of active drug.

It is planned to enroll more than or equal to 24 subjects with COVID-19. It is expected to have at least 12 evaluable patients in each group.

Experimental group: 0.4 mg/kg rhACE2 IV BID and standard of care Control group: standard of care

Intervention duration: up to 7 days of therapy

No planned interim analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Laboratory diagnosis:

   * Respiratory specimen is positive for SARS-CoV-2 nucleic acid by RT-PCR; OR,
   * The viral gene sequencing of the respiratory specimen is highly homologous to known novel coronavirus.
2. Fever:

   Axillary temperature >37.3℃
3. Respiratory variables (meets one of the following criteria):

   * Respiratory rate: RR ≥25 breaths/min
   * Oxygen saturation ≤93% at rest on room air
   * PaO2/FiO2 ≤300 mmHg（1 mmHg=0.133 KPa）
   * Pulmonary imaging showed that the lesions progressed more than 50% within 24-48 hours, and the patients were managed as severe
4. HBsAg negative, or HBV DNA ≤10^4 copy/ml if HBsAg positive; anti-HCV negative; HIV negative two weeks prior to signed Informed Consent Form (ICF)
5. Appropriate ethics approval and
6. ICF

Exclusion Criteria:

* Age <18 years; Age >80 years
* Pregnant or breast feeding woman or with positive pregnancy test result
* P/F <100 mmHg
* Moribund condition (death likely in days) or not expected to survive for >7 days
* Refusal by attending MD
* Not hemodynamically stable in the preceding 4 hours (MAP ≤65 mmHg, or SAP <90 mmHg, DAP <60 mmHg, vasoactive agents are required)
* Patient on invasive mechanical ventilation or ECMO
* Patient in other therapeutic clinical trial within 30 days before ICF
* Receive any other ACE inhibitors (ACEI), angiotensin-receptor blockers (ARB) treatment within 7 days before ICF
* Chronic immunosuppression: current autoimmune diseases or patients who received immunotherapy within 30 days before ICF
* Hematologic malignancy (lymphoma, leukemia, multiple myeloma)
* Other patient characteristics (not thought to be related to underlying COVID-19) that portend a very poor prognosis (e.g, severe liver failure, and ect)
* Known allergy to study drug or its ingredients related to renin-angiotensin system (RAS), or frequent and/or severe allergic reactions with multiple medications
* Other uncontrolled diseases, as judged by investigators
* Body weight ≥85 kg

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Time course of body temperature (fever) | 14 days
  Compare the time course of body temperature (fever) between two groups over time.
Viral load over time | 14 days
  Compare viral load between two groups over time.

SECONDARY OUTCOMES:
P/F ratio over time | 14 days
  PaO2/FiO2 ratio
Sequential organ failure assessment score(SOFA score) over time | 14 days
  SOFA, including assessment of respiratory, blood, liver, circulatory, nerve, kidney, from 0 to 4 scores in each systems, the higher scores mean a worse outcome.
Pulmonary Severity Index (PSI) | 14 days
Image examination of chest over time | 14 days
  Based on radiologist's assessment of inflammatory exudative disease, category as follows: significant improvement, partial improvement, no improvement, increase of partial exudation, significant increase in exudation, unable to judge.
Proportion of subjects who progressed to critical illness or death | 14 days
Time from first dose to conversion to normal or mild pneumonia | 14 days
T-lymphocyte counts over time | 14 days
C-reactive protein levels over time | 14 days
Angiotensin II (Ang II) changes over time | 14 days
Angiotensin 1-7 (Ang 1-7) changes over time | 14 days
Angiotensin 1-5 (Ang 1-5) changes over time | 14 days
Renin changes over time | 14 days
Aldosterone changes over time | 14 days
Angiotensin-converting enzyme (ACE) changes over time | 14 days
Angiotensin-converting enzyme 2 (ACE2) changes over time | 14 days
Interleukin 6 (IL-6) changes over time | 14 days
Interleukin 8 (IL-8) changes over time | 14 days
Soluble tumor necrosis factor receptor type II (sTNFrII) changes over time | 14 days
Plasminogen activator inhibitor type-1 (PAI-1) changes over time | 14 days
Von willebrand factor (vWF) changes over time | 14 days
Tumor necrosis factor-α (TNF-α) changes over time | 14 days
Soluble receptor for advanced glycation end products (sRAGE) changes over time | 14 days
Surfactant protein-D (SP-D) changes over time | 14 days
Angiopoietin-2 changes over time | 14 days
Frequency of adverse events and severe adverse events | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Yimin Li, PhD, MD, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- GCP Office of The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Zhang X, Li S, Niu S. ACE2 and COVID-19 and the resulting ARDS. Postgrad Med J. 2020 Jul;96(1137):403-407. doi: 10.1136/postgradmedj-2020-137935. Epub 2020 Jun 10. PMID 32522846